CLINICAL TRIAL: NCT01717092
Title: Epidemiological Study of Chronic Thromboembolic Pulmonary Hypertension in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Shengqing Li, MD, PhD, Associate Chief Physician, Associate Professor, Air Force Military Medical University, China
Other Study IDs: XJ-CTPH20121026
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: To Assess the Long-term Risk for Adverse Events After PE.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Consecutive patients with acute PE

SUMMARY:
Chronic thromboembolic pulmonary hypertension (CTPH) is associated with considerable morbidity and mortality. Its incidence after pulmonary embolism and associated risk factors are not well documented in Chinese population. We conducted a prospective, long-term, follow-up study to assess the incidence of symptomatic CTPH in consecutive patients with an acute episode of pulmonary embolism but without prior venous thromboembolism. Patients with unexplained persistent dyspnea during follow-up underwent transthoracic echocardiography and, if supportive findings were present, ventilation-perfusion lung scanning and pulmonary angiography. CTPH was considered to be present if systolic and mean pulmonary-artery pressures exceeded 40 mm Hg and 25 mm Hg, respectively; pulmonary-capillary wedge pressure was normal; and there was angiographic evidence of disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an episode of acute symptomatic pulmonary embolism without prior pulmonary embolism or venous thrombosis

Exclusion Criteria:

* Have other diseases (e.g., systemic sclerosis or severe emphysema) that could have caused nonthromboembolic pulmonary hypertension,
* Have preexisting exertional dyspnea,
* Geographically inaccessible for follow-up,
* Decline to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with an acute episode of pulmonary embolism but without prior venous thromboembolism.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
The cumulative incidence of symptomatic CTEPH | 2 years

SECONDARY OUTCOMES:
Risk factors for Recurrent VTE and CTEPH | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tangdu hospital, Xi'an, Shaanxi
  - Xijing hospital, Xi'an, Shaanxi